CLINICAL TRIAL: NCT01854177
Title: Differentiating the Effects of Substance P and Beta-endorphin in the Perception of Breathlessness During Resistive Load Breathing in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Differentiating the Effects of Substance P and Beta-endorphin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Donald A. Mahler, Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CPHS#23992
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: breathlessness; substance P; beta-endorphin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant (Active Comparator): Aprepitant 125 mg
  Interventions: Drug: Aprepitant
- Placebo (Placebo Comparator): Inert capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant
  Other Names: aprepitant 125 mg capsule
  Arms: Aprepitant
Drug: Placebo
  Other Names: inert capsule
  Arms: Placebo

SUMMARY:
In previous studies we demonstrated that endogenous opioids (inhibitory neuropeptides) modulate the perception of breathing difficulty in patients with chronic obstructive pulmonary disease (COPD). Recently, we found that antagonism of substance P (an excitatory neuropeptide) with aprepitant did not affect the perception of breathing difficulty. However, after administration of aprepitant, blood levels of both substance P(+ 54 ± 39%) and beta-endorphin (+ 27 ± 17%) increased significantly. As these blood levels reflect cellular/tissue activity, we postulated that the concomitant release of excitatory (substance P) and inhibitory (beta-endorphin) neuropeptides had opposing effects (counterbalanced each other) on the perception of breathing difficulty.

The objective of the present study is to further examine the possible role of substance P on the perception of breathlessness. We propose to administer oral aprepitant and oral placebo in a randomized clinical trial in patients with COPD. However, four hours after patients take these medications, intravenous naloxone will be administered in order to block the effects of endogenous opioids (beta-endorphin) on opioid receptors. Five minutes later, patients will breathe thru a tube with fine wire mesh to provoke breathing difficulty, and then provide ratings of the intensity and unpleasantness of breathlessness every minute.

The two competing hypothesis of the study are:

1. if breathlessness ratings with aprepitant/naloxone = placebo/naloxone, then substance P has no effect on perception of breathing difficulty;
2. if breathlessness ratings with aprepitant/naloxone ≠ placebo/naloxone, then substance P has an effect on perception of breathing difficulty.

DETAILED DESCRIPTION:
This study is a randomized, controlled clinical trial comparing the acute effects of oral aprepitant (selective antagonist of substance P receptor) vs. placebo on ratings of breathlessness during resistive load breathing in patients with COPD. Four hours after randomization, all patients will receive intravenous naloxone (antagonist of opioid receptors) to block the effects of endogenous opioids on perception of breathlessness. The two competing hypothesis of the study are:

Breathing difficulty will be induced by the patient breathing thru a tube with fine wire mesh for approximately 10 - 20 minutes in the laboratory.

Approximately 20 patients with COPD will be recruited from the out-patient clinic at the Dartmouth-Hitchcock Medical Center. The population will consist of female or male adults at least 50 years of age, at least 10 pack-year history of smoking, and a diagnosis of COPD associated with chronic bronchitis based on standard criteria.

ELIGIBILITY:
Inclusion Criteria:

* male or female patient 50 years of age or older
* a diagnosis of COPD; former smoker with a history of greater than or equal to 10 pack-years
* a clinical diagnosis of chronic bronchitis (productive cough on most days for a minimum of three months per year for at least two successive years)
* a post-bronchodilator forced expiratory volume in one second (FEV1) greater than or equal to 30% predicted and less than or equal to 80% predicted
* a post-bronchodilator FEV1/forced vital capacity (FVC) ratio less than 70%; and clinically stable COPD.

Exclusion Criteria:

* current smoker
* pregnant women
* current or previous (within the past two weeks) use or of a narcotic medication
* any patient who has a concomitant disease that might interfere with study procedures or evaluation including lactose intolerance
* use of a drug that may cause possible drug interaction with aprepitant [including cilostazol, dofetilide, ergot alkaloids, oral or non-oral contraceptives, progestins, ranolazine, reboxetine, warfarin, ziprasidone, anxiolytic medications, anti-depressive medications, cholesterol lowering drugs (e.g., atorvastatin, simvastatin), theophylline, antifungal antibiotics, and macrolide antibiotics]
* use of a contraindicated medication including astemizole, cisapride, pimozide, and terfenadine;
* use of angiotensin converting enzyme inhibitor

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald A Mahler, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study Population: Participants who consented and received both Aprepitant 125 mg taken orally and Placebo (Inert capsule taken orally) in random order 2-3 days apart.
Period: Overall Study
Arm/Group | Overall Study Population
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One patient was excluded from analysis because there was a 28% difference in her post-bronchodilator FEV1 between visits 2 and 3.
Groups:
- Entire Study Population: Includes groups randomized to receive Aprepitant first and placebo
Arm/Group | Entire Study Population
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Unpleasantness of Breathlessness
Description: Unpleasantness of breathlessness was reported each minute by the patient on a visual analog scale. The scale range is 0-10 where 0 = No breathlessness and 10 = Severe breathlessness. The measures were collected up to 20 minutes per visit and combined for a final score. Total minimum score = 0, total maximum score 200. Data is collected during Resistive Load Breathing at Period 1 (Day 3 or 4) and Period 2 (Day 5, 6 or 7) during which either Placebo or Aprepitant was administered. A high unpleasantness indicates that breathing difficulty feels very bad or terrifying regardless of whether the intensity is high or low
Time Frame: Visit 2 (Approximately Day 3 where either Placebo or Aprepitant was administered).and Visit 3 (approximately Day 6 where either Placebo or Aprepitant was administered)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Aprepitant: aprepitant 125 mg taken orally
- Placebo: inert capsule taken orally
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | 69.0 (24.9) | 71.1 (24.6)

2. Primary Outcome: Intensity of Breathlessness
Description: Intensity of Breathlessness was recorded on a visual analog scale. The scale range is 0-10 where 0 = minimum and 10 = maximal intensity. At each visit, participants were asked to report unpleasantness at 1 minute intervals. The measures were collected up to 20 minutes per visit and combined for a final score. Total minimum score = 0, total maximum score 200. Data is collected during Resistive Load Breathing at Period 1 (Day 3 or 4) and Period 2 (Day 5, 6 or 7) during which either Placebo or Aprepitant was administered.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | 83.0 (23.6) | 85.1 (20.5)

ADVERSE EVENTS:
Arm/Group | Aprepitant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Study assessed acute effects of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes